CLINICAL TRIAL: NCT02234778
Title: Evaluation of the Use of the Tissue Genesis® Icellator Cell Isolation System™ for Autologous Adipose-Derived Stromal Vascular Fraction Cells to Treat Critical Limb Ischemia
Brief Title: Evaluation of the Tissue Genesis® Icellator Cell Isolation System™ to Treat Critical Limb Ischemia
Acronym: CLI-DI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tissue Genesis (Industry)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TGI-002-01-2013
Record Dates: First submitted 2014-09-04; First posted 2014-09-09 (Estimated); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Critical Limb Ischemia
Keywords: critical limb ischemia; autologous stromal vascular fraction
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Treatment (Experimental): Each subject will receive up to 30 cc of the TGI SVF material via intramuscular injection (injections at multiple locations on the lower leg - up to 20 total injections) through a 23 gauge needle over a 2- to 4- minute period. TGI SVF material injection will be completed within 4 hours of cell separation.
  Interventions: Device: TGI SVF material via intramuscular injection

INTERVENTIONS:
Device: TGI SVF material via intramuscular injection — Each SVF-treated subject will receive up to 30 cc of the TGI SVF material via intramuscular injection (injections at multiple locations on the lower leg - up to 20 total injections) through a 23 gauge needle over a 2- to 4- minute period.

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of the Tissue Genesis® Icellator Cell Isolation System™ in Critical Limb Ischemia. The Icellator System™ device removes certain cells from the adipose (fat) tissue which will be used to treat patients with blockages in the arteries of their lower legs that may require a future amputation, which is caused by severe peripheral artery disease (PAD). The purpose of this study is to determine if treatment with cells that have been removed from the Icellator System™ device will reduce the number of major amputations and deaths in a six month time period.

ELIGIBILITY:
Inclusion Criteria:

* Critical limb ischemia (CLI), defined as ischemic pain at rest (Rutherford Category 4) or minor tissue loss of the limb (Rutherford Category 5), and with either toe artery occlusive pressure < 50 mmHg or TBI ≤ 0.5 or ankle artery occlusion pressure ≤ 60 mm Hg or ABI ≤ 0.5
* No reasonable open or endovascular surgical options as determined by treating vascular specialist
* Competent to give consent
* Age 21 years or greater
* Females of child bearing potential agree to use acceptable methods of contraception for the duration of the trial. Sexually active males agree to use an accepted and effective method of contraception for the duration of the trial.
* All diabetic subjects will undergo baseline and 12-month follow-up retinal examinations conducted by a specialist
* No current malignancy or history of previous malignancy within the last five years, with the exception of adequately treated non-melanoma cutaneous carcinoma (basal cell or squamous cell carcinoma of the skin).

Exclusion Criteria:

* Major tissue loss of the index limb (Rutherford Category 6)
* Limb revascularization surgery within 45 days of enrollment in this study
* Subjects with less than 15% body fat as measured by calipers or electrical impedance
* Subjects with less than a 2 cm x 2 cm roll of subcutaneous abdominal fat, when pinched between the examiner's fingers, while the subject is in a supine position
* Poorly controlled diabetes mellitus evidenced by HbA1C > 10%. Diabetic subjects must have evidence of a glycosylated hemoglobin test (HbA1C) performed within the last 30 days.
* Uncompensated congestive heart failure (New York Heart Association Class IV) and/or other conditions that preclude general anesthesia.
* Myocardial infarction or stroke within the last 90 days.
* Elevated liver function tests (AST or ALT more than twice the upper limit of normal).
* Hematologic abnormalities.
* Disease of the central nervous system and/or other conditions that impair cognitive function.
* History of two or more episodes of pulmonary embolus with a documented deep venous thrombosis (DVT) (Duplex US or venography) in the index extremity or history of DVT in the index extremity without evidence of clot resolution (Duplex US or venography)
* Infection of the index leg
* Pregnant or lactating females. Prior to enrollment, women of child-bearing potential must have a negative urine pregnancy test.
* Lower extremity venous disease or lymphedema with pitting edema in the index leg
* Osteomyelitis in the index leg
* Existing HIV diagnosis
* Known terminal disease process with a life expectancy of less than one year
* Subjects, in the investigator's opinion, requiring amputation within 30 days
* Uncorrected stenosis(es) of greater than 50% in the common and/or external iliac artery and/or common femoral artery of the index leg
* Presence of any clinical condition that in the opinion of the PI or the sponsor makes the patient not suitable to participate in the trial

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-08 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Amputation-Free Survival | 26 weeks
  To obtain preliminary feasibility evidence of the ability of the Tissue Genesis Inc. (TGI) stromal vascular fraction (SVF) material to result in freedom from major amputation (above the ankle) or death at 26 weeks following treatment. Treatment failure is defined as the composite of major amputation of the treatment limb or all-cause death.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States